CLINICAL TRIAL: NCT03164889
Title: Clinical and Basic Research of Relationship Between Hepatitis B Virus Quasi-Species Evolution and Function of Natural Killer Cells With Antiviral Therapy Response in Chronic Hepatitis B Patients
Brief Title: Clinical and Basic Research of ETV Plus GM-CSF in Chronic Hepatitis B Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no enough participant can be enrolled
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 首发2014-2-5033
Record Dates: First submitted 2016-11-15; First posted 2017-05-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2017-01

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B, antiviral treatment
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETV+GM-CSF (Experimental): Entecavir (ETV) plus Granulocyte Macrophage-colony Stimulating Factor (GM-CSF). ETV was given 0.5mg/d, oral; GM-CSF was given 100ug, the 3th, 4th, 5th day at week1, 4, 12, 24, 48, subcutaneous injection.
  Interventions: Drug: Granulocyte Macrophage-colony Stimulating Factor; Drug: Entecavir
- ETV monotherapy (Active Comparator): As standard antiviral therapy, Entecavir was given 0.5mg/d, oral.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Granulocyte Macrophage-colony Stimulating Factor — The intervention drug was used as an immunomodulator in order to improve rates of HBsAg loss and HBeAg loss.
  Other Names: GM-CSF
  Arms: ETV+GM-CSF
Drug: Entecavir — Antiviral drug for hepatitis b virus (HBV)
  Other Names: ETV

SUMMARY:
Previous studies indicated that Granulocyte Macrophage-colony Stimulating Factor (GM-CSF) could improve survival rate in patients with acute liver failure and obtain higher HBsAg seroconversion rate when in combination with peg-interferon for chronic hepatitis B (CHB) patients. In this study, investigators will study the clinical effect of entecavir (ETV) plus GM-CSF in patients with CHB compared to ETV monotherapy.

DETAILED DESCRIPTION:
Antiviral treatment plays critical role in treatment of chronic HBV infection. Entecavir, an nucleos(t)ide analogs (NA) targeting the viral polymerase, is widely used in China as the first line drug in antiviral treatment for CHB patients. The sustained suppression of serum HBV DNA to undetectable level has been proven to be associated with the prevention of progression of liver disease and inhibition of the development of hepatocellular carcinoma. According to data published, a rate about 70% HBVDNA undetectable could be reached after 1 year therapy. However, the rate of HBsAg loss is very low about 0% to 1%. Granulocyte-macrophage colony-stimulating factor(GM-CSF) is an important cytokine for the generation and propagation of antigen-presenting cells and for priming a cellular immune response. It increases the production of macrophage precursors and, in turn,enhances the T-helper cell (Th cell)-mediated cytotoxicity and regulates the tumoricidal cytokines. Previous studies indicated that when combined with IFN in patients with chronic HBV infection, it increased the therapeutic efficacy of the latter. Recent studies showed that GM-CSF benefit patients with acute liver failure. In this study, entecavir (ETV) plus GM-CSF would be used in patients with CHB compared to ETV monotherapy. Primary objective of the study is to see if there is significant improvement in HBsAg loss, rates of HBeAg loss and HBV undetectable are also to be observed. Function of NK cell from the patients enrolled will be measured during the therapy.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for more than 6 months
* HBeAg positive
* ALT≥80U/L or inflammation score ≥2 of histological examination

Exclusion Criteria:

* History of drug allergy to GM-CSF
* coinfection with HCV, HIV, HAV, HEV
* liver cirrhosis or CHILD score >7
* diagnosis of hepatocellular carcinoma or AFP>100ng/ml
* Allergic thrombocytopenic purpura

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of HBsAg loss | 48 weeks after therapy

SECONDARY OUTCOMES:
Rate of HBeAg loss | 48 weeks after therapy
HBVDNA undetectable rate | 48 weeks after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ping Zhao, Director, Study Director — 302 Military Hospital, Beijing, China
Locations (1):
- 302 Military Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No